CLINICAL TRIAL: NCT06226259
Title: Improvement Effects of Gamma Aminobutyric Acid（GABA） Supplementation on Treatment of Children With Insomnia, A Randomized, Placebo-controlled, Single-center, Intervention Study
Brief Title: Improvement Effects of Gamma Aminobutyric Acid（GABA） Supplementation on Treatment of Children With Insomnia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Guanghai Wang, Principal Investigator，Professor, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LY202330154
Record Dates: First submitted 2023-12-26; First posted 2024-01-26 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GABA supplement group (Experimental): The experimental group was given a kind of GABA supplement already on the market, with 100mg of GABA in the unit package.
  Take orally every night before sleep for 14 days.
  Interventions: Dietary Supplement: GABA supplement
- placebo group (Placebo Comparator): Placebo ,Take orally every night before sleep for 14 days.
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: GABA supplement — Oral administration of GABA supplement once daily before sleep for 14 days.
  Arms: GABA supplement group
Dietary Supplement: placebo — Oral administration of placebo once daily before sleep for 14 days.
  Arms: placebo group

SUMMARY:
Around 20% of children worldwide suffer from insomnia. There are no approved drugs available for treating insomnia in children, and there may be treatment-related side effects. The Gamma aminobutyric Acid (GABA) is a neurotransmitter widely present in the brain, and GABA extracted by industry is a common food supplement. Previous studies indicate that oral GABA supplement can improve adult insomnia, and has the potential to reduce blood pressure, relieve stress and other effects. At present, there are few studies using oral GABA to improve insomnia in children. The purpose of the study is to explore the effects of oral GABA supplement on symptoms of insomnia (short - or long-term insomnia) in children. In this study, 206 children aged 6-12 years with a diagnosis of insomnia will be randomly assigned to receive GABA supplement of 100mg/ day or placebo for 2 weeks. Subjective and objective sleep parameters such as sleep onset latency (SOL) were measured with sleep questionnaires, diary, and actigraphy at baseline and 2 weeks later, while emotional/behavioral problems, and cognitive ability will be measured with parent-reported questionnaires. Also, related brain function was assessed with functional near-infrared spectroscopy (fNIRS). This study can provide more reference for the application of GABA in children with insomnia as a complementary and alternative therapy, and clarify the mechanism of action of GABA on insomnia.

DETAILED DESCRIPTION:
Children aged 6-12 years with insomnia will be randomly assigned to GABA supplement group and placebo group in a 1:1 ratio. Participants will be provided with corresponding interventions. The experiment group was given a common food GABA supplement already on the market, with 100 mg of GABA in the unit package. The placebo group replaced the equivalent amount of GABA with a placebo component of starch. Placebo and GABA supplement are identical in appearance to guarantee blindness. Subjects will be followed up at baseline and 2 weeks after taking the test supplementary GABA to assess its effect on symptoms of insomnia, psychological and emotional status, and as well as related brain functions.

All questionnaires will be filled out by the primary caregivers, and the physical examination data will be measured at Shanghai Children's Medical Center. Information on insomnia diagnosis, disease classification, current treatment, and comorbidities will be obtained from daily medical visit records.

This study was a randomized double-blind controlled trial. All participants in the study will be divided into two groups: GABA supplement in the intervention group and placebo in the control group. Both groups will be provided education of sleep hygiene. Participants should take GABA supplements or placebo once daily before sleep for 14 days. The primary endpoint is the change in sleep onset latency (SOL) from baseline at two weeks after the trial as assessed by sleep dairy and actigraphy. Secondary assessment indicators: Total sleep time（TST）; Sleep efficiency(SE); Wake after sleep onset(WASO); Time in bed(TIB); Children's Sleep Habits Questionnaire(CSHQ) . Changes of children's emotional and cognitive functions before and after intervention will be assessed using functional near-infrared spectroscopy（fNIRS） and relevant psychological scales . Adverse events(AE) will be closely monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Children （both male and female）age 6-12 years
* Clearly diagnosed as chronic or short-term insomnia according International classification of sleep disorders-third edition（ICSD-3）
* No hearing or vision impairment, able to follow simple instructions from clinicians or parents
* Have not participated in any drug clinical trials within 3 months at the screening point
* The child or family member has the ability to evaluate and fill in a sleep diary and operate an actigraphy
* Sign informed consent

Exclusion Criteria:

* Previously diagnosed and known to be associated with intellectual disability (IQ ≤ 70)
* Clear diagnosis of anxiety disorder in the past
* Clear diagnosis of depression
* Suffering from serious cardiopulmonary and blood system diseases, low immune function, and physical diseases
* Suffering from mental developmental disorders associated with sleep disturbance and major psychosis, including well-defined (autism spectrum disorder; Attention deficit hyperactivity disorder; Schizophrenia; Schizoaffective disorder; Bipolar disorder;Post-traumatic stress disorder; Compulsive disorder; Mental disorders caused by epilepsy etc.)
* Suffering from other disorders associated with insomnia, including well-defined diagnoses (sleep apnea, periodic limb movement disorder, restless leg syndrome and nocturnal frontal lobe epilepsy, circadian dysrhythmia sleep disorder)
* Use of drugs that affect sleep (e.g. sleeping pills, sedatives, antiasthmatics, melatonin, antihistamines)
* Suffering from allergies or allergies to milk proteins and lactose intolerance
* The researchers think that is not suitable for other conditions (for example: nearly three months in other clinical research and are taking any other intervening drugs)
* Informed consent could not be obtained

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 206 (Estimated)
Dates: Start 2024-03-25 (Actual); Primary Completion 2025-11-12 (Estimated); Study Completion 2025-12-22 (Estimated)

PRIMARY OUTCOMES:
Change of sleep onset latency (SOL) of actigraphy | Baseline, Week 2
  sleep onset latency (minutes)

SECONDARY OUTCOMES:
Change of total sleep time （TST）of actigraphy | Baseline, Week 2
  total sleep time(minutes)
Change of sleep efficiency(SE) of actigraphy | Baseline, Week 2
  sleep efficiency (%)
Change of wake-time after sleep onset (WASO)of actigraphy | Baseline, Week 2
  wake-time after sleep onset (minutes)
Change of time in bed (TIB) of actigraphy | Baseline, Week 2
  time in bed (minutes)
Children's Sleep Habits Questionnaire （CSHQ） | Baseline, Week 2
  A quantitative scale used to assess sleep habits in children,the CSHQ consists of 33 items. The instrument evaluates the child's sleep based on behavior within eight different subscales: bedtime resistance, sleep-onset delay, sleep duration, sleep anxiety, night wakings, parasomnias, sleep-disordered breathing, and daytime sleepiness.
  Each item can be rated 1 -3，some items（item 1,2,3,10,11，26） need to be scored in reverse due to language representation. The cumulative total score is 33 - 66, The higher the score on the scale, the more poor the sleep habit.
insomnia symptoms:Athens Insomnia Scale (AIS) | Baseline, Week 2
  The Athens Insomnia Scale (AIS) measures severity of insomnia symptoms. The cumulative total score is 0-24;The total scores of these questionnaires were interpreted as follows: normal (0-6), mild (7-9), moderate (10-15), severe (16-24)insomnia.
Child sleep diary | Baseline, Week 2
  Parent-report child's sleep diary will be collected. Sleep parameters include bedtime, wake time, total sleep time, sleep onset latency, wake time after sleep onset, and the number of awakenings.
Griffith Empathy Measure Score | Baseline, Week 2
  Griffith Empathy Measure (GEM ), is a 23-item parent-report measure of affective and cognitive empathy. The maximum score is 92. Higher scores reflect higher reported empathy.
Child emotion:The Chinese Version of Spence Children's Anxiety Scale-Short Version | Baseline, Week 2
  This scale is used to assess anxiety in children which is a four-point Likert scale, from 0(never) to 3(always).The cumulative total score is 0-57 ,the higher the score, The more severe the anxiety.
Child emotion:Center for Epidemiologic Studies Depression Scale for Children (CES-DC) | Baseline, Week 2
  CES-DC is a self-rated depression questionnaire composed of 20 self-rated items with a total score ranging from 0 to 60 points, the higher the score, the higher the level of depression. The cutoff is 15 , scores above 15 indicating that depressive symptoms have a significant standard.
Executive Function | Baseline, Week 2
  Behavior Rating Inventory of Executive Function(BRIEF) is designed to assess executive function behaviors of children and adolescents aged 5-18 years in the home and school environments. It includes 86 items which divided 8 dimensions. The score will be converted to T score.When the Global Executive Composite or one of the 8 dimensions T score come to 65,impaired executive function should be considered.Higher scores represent poorer executive function.
Child neuro-changes | Baseline, Week 2
  The functional near-infrared spectroscopy (fNIRS) can collect the oxygenated hemoglobin and deoxyhemoglobin during brain activity.

OTHER OUTCOMES:
Parental emotion:Generalized Anxiety Disorder-7(GAD-7) | Baseline, Week 2
  The GAD-7 scale is a 7-item measure. The total score indicates anxiety severity over the last two weeks.
  The total scores of these questionnaires were interpreted as follows:range 0-21， normal (0-4), mild (5-9), moderate (10-14), and severe (15-21) anxiety.
Parental emotion:Patient Health Questionnaire-9(PHQ-9) | Baseline, Week 2
  The PHQ-9 is a 9 item measure. range: 0-27，The total score indicates severity of depression over the last two weeks.The total scores of these questionnaires were interpreted as follows: normal (0-4), mild (5-9), moderate (10-14), and severe (15-27) depression.
Parental life quality | Baseline, Week 2
  World Health Organization Five-item Well-Being Index(WHO-5),Range 0-25,the higher score the happier life,the cutoff is 13.
Parental sleep | Baseline, Week 2
  Pittsburgh Sleep Quality Index (PSQI)，total score range between 0 and 21,with higher numbers representing worse sleep quality
Parental satisfaction | Week 2
  A five-point Likert scale will be used to assess marital satisfaction. Scores range from 0 to 20. Higher scores reflect better marital satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Children's Medical Center, School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China